CLINICAL TRIAL: NCT07249073
Title: Exploratory Clinical Study on the Safety and Efficacy of CAR19-BCMA Dual-target CAR-T in the Treatment of Relapsed / Refractory Multiple Myeloma
Brief Title: CAR19-BCMA Dual-target CAR-T in the Treatment of Relapsed / Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025040
Record Dates: First submitted 2025-07-31; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR19-BCMA CAR-T (Experimental): This part follows the "3+3" dose escalation mode, with three dose groups (1E+06, 2E+06 and 3E+06 CAR+ cells /kg)
  Interventions: Drug: CAR19-BCMA dual-target CAR-T

INTERVENTIONS:
Drug: CAR19-BCMA dual-target CAR-T — This drug is CAR-T cell injection. CAR-T cells are based on the traditional CAR-T treatment, using cytokine combination amplification and improved transfection technology to change the activation mode of T cells.

SUMMARY:
1. Objective to evaluate the safety and tolerability of CAR19-BCMA dual-target CAR-T in the treatment of relapsed / refractory multiple myeloma.
2. To determine the maximum tolerated dose (MTD) of car19-bcma dual target car-t in the treatment of relapsed / refractory multiple myeloma.

DETAILED DESCRIPTION:
This study is an open, single arm, prospective, phase I clinical study, using "3+3" dose escalation to explore the safety, maximum tolerated dose, in vivo pharmacokinetic characteristics and preliminary efficacy of CAR19-BCMA dual-target CAR-T cell injection in the treatment of relapsed / refractory multiple myeloma subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all the following criteria to be enrolled in the study:

1. With Subjects' consent and signed informed consent, Subjects are willing and able to follow the planned visit, study treatment, laboratory examination and other test procedures; 2. Patients with relapsed / refractory multiple myeloma according to clinical diagnosis:

1. The expression of BCMA and / or CD19 in myeloma cells was positive confimed by flow cytometry or immunohistochemistry;
2. Patients with relapsed / refractory multiple myeloma who have received at least 1 line treatment (including proteasome inhibitors (PI), immunomodulatory drugs (IMID), CD38 mAb) or are resistant to proteasome inhibitors and / or immunomodulatory agents and / or CD38 mAb in the past.

3. Age 18-70 years old, both male and female; 4. Subjects with physical fitness status of 0-2 in the Eastern Cooperative Oncology Group (ECOG) score; 5. The estimated survival time from the date of signing informed consent is more than 3 months; 6. Hgb ≥ 60g/L (transfusible); 7. Liver and kidney function and cardiopulmonary function meet the following requirements:

1. Creatinine ≤ 2 × ULN;
2. Left ventricular ejection fraction ≥ 50%;
3. Blood oxygen saturation >90%;
4. Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN; 8. Subjects with pregnancy plans must agree to take contraception before enrollment in the study and after six months of study duration; The investigator should be informed immediately if the subject is pregnant or suspected of pregnancy.

   -

   Exclusion Criteria:

   If any of the following criteria is met, you cannot be enrolled:

   1. There were severe cardiac insufficiency and left ventricular ejection fraction <50%; 2. Have a history of severe lung function impairment disease; 3. Combined with other advanced malignant tumors; 4. It was complicated with serious infection and could not be effectively controlled; 5. Complicated with severe autoimmune disease or innate immune deficiency; 6. Active hepatitis (hepatitis B virus deoxyribonucleic acid [hbv-dna] or hepatitis C virus ribonucleic acid [hcv-rna] test results are higher than the lower limit of detection); 7. Human immunodeficiency virus (HIV) infection or known acquired immune deficiency syndrome (AIDS), or syphilis infection; 8. Have a history of severe allergy to biological products (including antibiotics); 9. One month after immunosuppressant withdrawal, patients with acute graft-versus-host response (GVHD) after allogeneic hematopoietic stem cell transplantation still exist; 10. There are other serious physical or mental diseases or abnormal laboratory tests that may increase the risk of participating in the study, or interfere with the results of the study, as well as patients who the investigator believes are not suitable for participating in this study; 11. Female patients (patients with fertility) are in pregnancy or lactation. Note: severe infection: refers to the infection with uncontrolled sepsis or infection focus, which can be enrolled after infection control.

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-03-27 (Estimated); Study Completion 2029-03-27 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | in 3 months after CART infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Laboratoty tests | in 3 months after CART infusion
  Abnormal results of laboratoty tests

SECONDARY OUTCOMES:
Overall response rate (ORR) | Day28, Month2, Month3, Month6, Month12, Month18, Month24 after CAR-T infusion
  Percentage of subjects who achieved minimal response (MR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigators
Minimal Residual Disease (MRD) negative rate | Day28, Month2, Month3, Month6, Month12, Month18, Month24 after CAR-T infusion
  Proportion of subjects who achieved MRD negative
Overall Survival (OS) | Minimum of 2 years post CAR-T infusion
  Time from CAR19-BCMA CAR-T infusion to time of death due to any cause
Progression-free Survival (PFS) | Minimum of 2 years post CAR-T infusion
  Time from CAR19-BCMA CAR-T infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first
Event-free Survival (EFS) | Minimum of 2 years post CAR-T infusion
  Time from CAR19-BCMA CAR-T infusion to time of disease progression, recurrence, death, etc
Disease Control Rate (DCR) | at Day28, Month2, Month3 , Month6, Month12, Month18, Month24 after CAR-T infusion
  disease control rate after CAR19-BCMA CAR-T infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xu, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China